CLINICAL TRIAL: NCT05328011
Title: Targeting Microbiota in Female Overactive Bladder Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Wolfgang Umek, MD, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Other Study IDs: 2160/2019
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Microbiota; Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- overactive bladder syndrome: female patients with overactive bladder syndrome
- controls: women without overactive bladder syndrome

SUMMARY:
The aim of this study is to compare the urinary viral microbiome and bacterial microbiome between overactive bladder syndrome (OAB) patients and healthy controls in order to determine a possible alteration in the urinary microbiome which may predispose women for OAB, and also in order to determine a possible influence of the urinary viral microbiome on the urinary bacterial microbiome which may predispose the individual to OAB. Furthermore, we aim to compare the urinary bacterial microbiome to the vaginal, rectal, urethral and salivary bacterial microbiome within the same individual and between the two groups in order to determine a possible route of colonization of the urinary bladder.

ELIGIBILITY:
Inclusion Criteria (case group):

* symptoms of overactive bladder (urgency with or without urinary leakage, usually with frequency and nocturia)

Exclusion Criteria (case group):

* Pregnant or lactating females

  * Neurological conditions (such as MS, Parkinson, spinal cord injury, stroke..)
  * Pelvic Organ Prolapse (stage ≥ 3)
  * Lower Urinary Tract surgery within past 6 months
  * Known history of interstitial cystitis or pain associated with OAB
  * Recurrent urinary tract infections > 3/year
  * Acute urinary tract infection
  * Urinary retention (with or without required self- catheterization)
  * Stress urinary incontinence or mixed urinary incontinence
  * Bladder cancer
  * Renal insufficiency
  * Urinary tract stones

Inclusion Criteria (control group):

without symptoms of overactive bladder or any other form of lower urinary tract symptoms

* Age-matched to case group (+/- 5 years)
* BMI-matched to case group (18,5- 24,9 kg/m2 normal weight; 25- 29,9 kg/m2 overweight; 30- 34,9 kg/m2 obesity grade I)

Exclusion criteria (control group):

As case group plus any form of lower urinary tract symptoms including OAB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients bothering for OAB, who present themselves at the urogynecological outpatient clinic, are considered to be eligible for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
urinary bacterial and viral microbiome | 1 day

SECONDARY OUTCOMES:
bacterial and viral microbiome of vagina, urethra, feces and oral cavity | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No